CLINICAL TRIAL: NCT00231855
Title: Phase II Trial- Weekly Taxotere and Topotecan for Recurrent Ovarian, Primary Peritoneal, Endometrial and Uterine Cancers
Brief Title: Efficacy Study of Weekly Taxotere and Topotecan for Recurrent Gynecologic (GYN) Cancers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Collaborators: Sanofi (Industry); GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Mark H. Einstein, Director, Clinical Research for Women's Health, Montefiore Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MMC-04-05-131
Record Dates: First submitted 2005-09-30; First posted 2005-10-04 (Estimated); Last update posted 2012-04-24 (Estimated); Status verified 2012-04

CONDITIONS: Ovarian Neoplasms; Uterine Neoplasms
Keywords: Epithelial Ovarian Cancer; Uterine Cancer; Prior Therapy; Chemotherapy; Recurrence
MeSH Terms: conditions — Ovarian Neoplasms; Uterine Neoplasms; Carcinoma, Ovarian Epithelial; Recurrence | interventions — Topotecan; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Topotecan and Taxotere

SUMMARY:
The primary aim of this study is:

* To determine the overall clinical response rate of weekly Topotecan and Taxotere in women with recurrent ovarian, primary peritoneal, endometrial and uterine cancers.

The secondary aims of this study are:

* To evaluate the safety and tolerability of the combination therapy with weekly Topotecan and Taxotere in patients with recurrent ovarian, primary peritoneal, endometrial or uterine cancers.
* To determine the progression free survival and overall survival in women treated with weekly Topotecan and Taxotere in patients with recurrent ovarian, primary peritoneal, endometrial and uterine cancers who have been previously treated with chemotherapy and/or radiation therapy.

DETAILED DESCRIPTION:
Endometrial carcinoma is the most common gynecologic cancer, accounting for 6,500 deaths in 2002 in the United States. There has been a 128% increase in endometrial cancer deaths over the past decade mainly due to recurrences. Although primary surgery with or without adjuvant therapy can cure most patients, effective therapy for those patients with advanced or recurrent disease is needed. Due to the advanced age of this patient population and associated medical comorbidities, these patients are not always ideal candidates for experimental therapies exploring dose intensity or toxic agents. Treatment options for advanced or recurrent disease are limited. Cytotoxic therapy has made little impact on survival.

Recent data has demonstrated efficacy of Topotecan in advanced or recurrent endometrial cancer. A Phase II trial performed primarily by the New York Gynecologic Oncology Group through ECOG found Topotecan to be an active first line treatment for metastatic or recurrent endometrial cancer. The overall response rate was 20% with 3/40 patients complete responders. A Phase II trial by the Gynecologic Oncology Group (GOG) of 29 patients with advanced or recurrent endometrial cancer reported a 10% overall response rate to 5-day intravenous Topotecan. However, 55% of patients had stable disease. Reported side effects were mainly hematologic, specifically, neutropenia and thrombocytopenia. Finkler and Holloway reported a phase I/II trial using weekly Topotecan in recurrent endometrial cancer. 23% of patients had partial response to therapy, with a decrease in grade 4 neutropenia and thrombocytopenia compared to the 5-day infusion. In a pilot study examining the role of 5-day Topotecan in uterine papillary serous carcinoma (UPSC), Chambers et al. report 11 of 12 patients who received Topotecan as front-line therapy to be disease-free at 13 months median follow-up. Anemia and neutropenia were managed effectively with hematopoietic stimulating factors.

Taxanes have also been reported to be effective in the treatment of advanced and recurrent endometrial cancer. Endometrial cancer cell lines have demonstrated sensitivity to paclitaxel. Response rates of 35%-37% have been reported in two separate phase II trials. Günthert et al., reported a complete response to Taxotere in a patient with recurrent endometrial cancer.

Taxotere is an agent well documented in the management of advanced ovarian cancer, with a response rate of approximately 30% in platinum-refractory patients. Taxotere has also demonstrated clinical response in patients classified as paclitaxel-refractory, confirming an incomplete cross-resistance between these two agents. Based on these data, there is reason to believe that the combination of Topotecan and Taxotere in the second-line setting may prove promising in patients initially treated with paclitaxel and platinum-based therapy.

Topotecan and Taxotere have known activity in ovarian cancer patients. Recent weekly dosing schedules suggest similar activity in ovarian cancer patients with less toxicity. Ovarian cancer patients who have significant Taxane-related side effects, including neuropathy, do well with weekly Taxotere. Both Topotecan and Taxotere have documented efficacy in recurrent endometrial cancer, but no study, to date, has utilized them in combination for the treatment of endometrial cancer. In addition to utilizing this regimen in a phase II setting for recurrent ovarian cancer, we propose a phase II trial utilizing this combination for the treatment of recurrent endometrial cancer. The justification for including all of these tumor types in the same protocol is the known similar response rates of these Gynecologic tumors to all chemotherapies. The endpoints and power are designed for all of the histologic types, but subset analysis will be used for each tumor type after completion of the trial.

Because of the broad spectrum of antitumor activity of both Topotecan and Taxotere, several phase I/II trials have been conducted with this combination regimen. Lu and colleagues at MD Anderson administered docetaxel (Taxotere) intravenously on Day 1 followed by bolus daily intravenous Topotecan on days 1-3 with subcutaneous Neupogen (Filgrastim) support on days 4-13. Dose limiting toxicity for the regimen was febrile neutropenia, and the recommended dose for phase II trials was docetaxel 75 mg/m2 IV on day 1 and topotecan 1.4 mg/m2 IV on days 1-3 with Neupogen (filgrastim) 5 mcg/kg/d SC on days 4-13. Three of the 11 patients enrolled experienced a response with the combination (1 CR and 1 PR in nasopharynx cancer and 1 PR in SCLC). Aijaz and colleagues at New York Medical Center conducted a similar pilot study in patients with recurrent ovarian and primary peritoneal cancer. In this trial, all of the patients received docetaxel 80 mg/m2 IV on day 1 and topotecan 1.0 mg/m2 IV on days 1-5. The patients also received Neupogen (filgrastim) 10-mcg/kg beginning on day 6 and continuing until the neutrophil count recovered to ≥ 10,000/mL. The regimen was relatively well tolerated, with neutropenia being the most frequently reported side effect. Preliminary antitumor activity was impressive, with 1 complete response, 4 partial responses, and 4 stable diseases reported among the twelve patients enrolled in the pilot study. A final phase I study combining topotecan and docetaxel was also conducted at The University of Wisconsin by Stella and colleagues. In this trial docetaxel was administered IV on day 1 followed by daily IV bolus Topotecan on days 1-5. In contrast to the previous studies, prophylactic growth factor support was not administered following chemotherapy administration. Because of significant myelosuppression at the initial dose level, the protocol was amended and the starting dose of Topotecan was reduced. As expected, the dose-limiting toxicity was myelosuppression consisting of both neutropenia and thrombocytopenia. The maximum tolerated dose for the combination regimen was docetaxel 60 mg/m2 IV on day 1 followed by Topotecan 0.75 mg/m2/d on days 1-5.

Recently, the combination of Topotecan and Taxotere has been used in a Phase I setting in platinum sensitive patients with recurrent ovarian and primary peritoneal cancers. Eleven patients have been treated to date with weekly docetaxel 30 mg/m2/wk plus topotecan 3.5 mg/m2/wk. Two patients were non-evaluable, one due to rapidly progressive disease and one due to noncompliance. Of the nine evaluable patients, five patients experienced dose-limiting toxicities as follows,

1. cycle 1 day 15 (C1D15) held due to platelets 33K in a heavily pretreated patient, including previous oxaliplatin,
2. C1D15 dose decreased due to grade 3 diarrhea,
3. C1D8 held due to grade 3-4 nausea and vomiting (may have been disease related),
4. C1D15 held due to platelets 49 K (74 yo, heavily pretreated including previous XRT),
5. C1D15 held due to platelets 43K and declining creatinine clearance of 43 ml/min (3 prior regimens, including XRT, PS 2 and history of thrombocytopenia).

One additional patient is planned to complete this dose level, to provide 10 evaluable patients. Of the 36 patients receiving 76 cycles of therapy, myelosuppression was brief and reversible with no febrile neutropenia. Per verbal communication from Dr. Burris, the recommended phase II dose will be docetaxel 30 mg/m2/wk plus topotecan 3.5 mg/m2/wk on days 1, 8 and 15 every 28 days for minimally pretreated patients.

In addition to possible synergy with this combination of drugs in other tumor types, the weekly dosing may have a better safety profile. The dose-limiting toxicity for Topotecan when administered on a daily x 5-administration schedule is myelosuppression. However, when the drug is administered on a weekly administration schedule, the myelosuppression is ameliorated and is no longer dose limiting. Additionally, weekly docetaxel administration is gaining in popularity in the clinical arena due to the improved toxicity profile of the drug. The possibility of synergy with the improved safety profile secondary to weekly dosing makes this combined dosing regimen a rational possibility for this patient population.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented recurrent endometrial adenocarcinoma, papillary serous (UPSC), or mixed mullerian tumor (MMT) for which a cure or substantial palliation is unlikely using surgery and/or radiotherapy. Patients must have measurable disease or disease felt to be reproducibly measurable on CT scan, chest x-ray and/or tumor marker elevations .
* Recurrent ovarian or primary peritoneal cancers as defined as either:

  1. Measurable disease either by physical examination or by imaging or
  2. Non-measurable evidence of disease such as any or all of the following standard Rustin criteria:

     1. Peritoneal implants <2 cm
     2. Abnormal densities on computerized tomography (CT) scan and/or loculated fluid collections
     3. Elevated CA-125 (>100 U/mL on 2 measurements at least 1 week apart) and disease- related symptoms.
* Patients with the following histologic ovarian or uterine epithelial cell types are eligible:

  * Serous adenocarcinoma
  * Endometrioid adenocarcinoma
  * Mucinous adenocarcinoma
  * Undifferentiated carcinoma
  * Clear cell adenocarcinoma
  * Mixed epithelial carcinoma
  * Transitional cell
  * Malignant Brenner's tumor
  * Adenocarcinoma NOS
* Age ≥ 18 years.
* ECOG performance status of ≤ 2.
* Peripheral neuropathy must be ≤ grade 1
* Previously treated patients must have received no antineoplastic treatment for at least 4 weeks. Patients will not have received more than two previous chemotherapy regimens.
* In patients previously irradiated, the recurrent disease should be outside of the radiotherapy portal or have developed disease progression within the radiated field.
* No concurrent chemotherapy, radiotherapy, immunotherapy, or hormone therapy.
* Hepatic:

  * Total bilirubin ≤ ULN
  * AST and ALT and alkaline phosphatase must be within the range allowing for eligibility.
* Patients must be alert, oriented, and have signed an informed consent in accordance with institutional policies and be aware of the investigational nature of the study.
* Women of childbearing potential must be willing to consent to using effective contraception while on treatment and for at least 3 months thereafter

Exclusion Criteria:

* Patient has impairment of hepatic, renal or hematologic function as defined by the following baseline laboratory values:

  1. Serum creatinine clearance ≤ 50 ml/min
  2. Platelets <100,000/mm3
  3. Absolute neutrophil count (ANC) <1500/mm3
  4. Hemoglobin <8.0 g/dl (the patient may be transfused prior to study entry)
* History of chronic or active hepatitis
* Patient has severe or uncontrolled medical disease (eg. uncontrolled diabetes, unstable angina, myocardial infarction within 6 months, congestive heart failure, etc.)
* Patients with dementia or altered mental status that would prohibit the giving and understanding of informed consent at time of study entry.
* Patients with a history of severe hypersensitivity to Taxotere®, Topotecan®, or other drugs formulated with polysorbate 80.
* Women who are pregnant or breast-feeding

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31
Dates: Start 2004-11; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
To determine the overall clinical response rate of weekly Topotecan and Taxotere in women with recurrent ovarian, primary peritoneal, endometrial and uterine cancers

SECONDARY OUTCOMES:
To evaluate the safety and tolerability of weekly Topotecan and Taxotere in patients with recurrent ovarian, primary peritoneal, endometrial or uterine cancers
To determine the progression free survival and overall survival with weekly Topotecan and Taxotere in patients with recurrent ovarian, primary peritoneal, endometrial and uterine cancers who have been previously treated with chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Mark H Einstein, M.D., M.S., Principal Investigator — Montefiore Medical Center and Albert Einstein College of Medicine
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

REFERENCES:
- [Result] Gupta D, Owers RL, Kim M, Kuo DY, Huang GS, Shahabi S, Goldberg GL, Einstein MH. A phase II study of weekly topotecan and docetaxel in heavily treated patients with recurrent uterine and ovarian cancers. Gynecol Oncol. 2009 Jun;113(3):327-30. doi: 10.1016/j.ygyno.2009.02.018. PMID 19307014